IRB – 16-1571 Consent Version 3/23/2020

# The Cleveland Clinic Foundation Consent to Participate in a Research Study

Study title: Efficacy of Exparel ® on Post-operative Pain after Laparoscopic Gastric Bypass

Using Circular EEA Stapler

Sponsor: Pacira Pharmaceuticals, Inc.

Principal Investigator: Dr. John Rodriguez, 216-445-9966

You are being invited to participate in a research study. A research study is designed to answer specific questions about new ways to prevent, detect, and treat disease. The purpose of this document is to provide a written summary of the discussion of research information you had with the research team to help you decide if you wish to participate in research. It is important for you to ask questions and understand the risks, benefits and alternatives.

#### Please note:

- You are being asked to participate in a research study
- Carefully consider the risks, benefits, and alternatives of the research
- Your decision to participate is completely voluntary

## 1. INFORMATION ON THE RESEARCH

### Why is the research study being done?

During an operation, a drug called Bupivacaine is routinely injected around an incision to decrease post-operative pain. Bupivacaine is approved by the United States Food and Drug Administration (FDA) for pain relief after surgery, and is the current standard of care.

A form of Bupivacaine that acts for a longer period of time, Liposomal Bupivacaine (Exparel®), is now available. This study will compare post-operative pain among patients undergoing laparoscopic gastric bypass who are either given Bupivacaine alone or in combination with Liposomal Bupivacaine (Exparel®).

This research will take place at the Cleveland Clinic. You are being asked to participate in this study because you are scheduled to have laparoscopic gastric bypass surgery.

#### How Many People Will Take Part In The Study?

About 100 people will take part in this study.

#### What Is Involved In The Study?

This is a blinded, randomized, control study. Randomized means that you will be selected (like flipping a coin) to one of the following treatment groups:

IRB – 16-1571 Consent Version 3/23/2020

- Control group: 60cc Bupivacaine
- Experimental group: 20cc Liposomal Bupivacaine (Exparel®) and 40cc Bupivacaine

Blinding means that you and the study staff that assess your pain control after your operation will not know which medication you received. However, in an emergency, the study team can quickly find out what group you are assigned to. If you are assigned to the control group, you will receive the current standard of care drug.

Prior to your operation: There will be no change to the preoperative evaluation and education process for your bariatric operation. A member of the study staff will review the study with you and you sign this consent form prior to your operation.

During your hospital stay: While you are in the operating room, the control or experimental drug will be injected around your incisions before you awake from general anesthesia. All other parts of your operation will be standard of care.

A member of the study team, who will not know what medication you received, will visit you while you are in the hospital to administer a questionnaire about your pain control. Your surgical team will monitor for occurrence of post-operative symptoms such as nausea, vomiting, infections, complications related to the surgery, and your body's reaction to the study drug. Information about the amount of other pain control medication you use will be gathered after you are discharged from the hospital.

Follow up visits after discharge from the hospital: There is a standard schedule for post-operative appointments after bariatric surgery. Your fist visit is 7-10 days after your hospital discharge. The purpose of this visit is to detect any early post-operative complications and to give you a chance to ask questions. The second visit is 1 month after surgery.

A timeline is below. Your participation in this study will last approximately 1 month after your operation.



IRB – 16-1571 Consent Version 3/23/2020

### 2. ALTERNATIVES

## What are the alternatives to participation in the research study?

The alternative to enrolling in this study is electing not to participate. You will still receive the standard post-operative pain control. Deciding not to participate will not affect your care now or in the future at Cleveland Clinic.

#### 3. RISKS

What are the risks of participating in the research study?

### **Unforeseeable-Unknown Risks:**

There may be risks or side effects related to the study medications that are unknown at this time. Any research has some risks, which may include things that could make you feel uncomfortable, or harm you. All research participants taking part in the study will be watched carefully for any negative effects. You will be notified of any significant new findings that become known that may affect your willingness to continue in the study.

### Possible risks of Bupivacaine:

Mild: Headache, insomnia (inability to fall asleep), muscle spasms (twitching), or back pain.

Moderate: Akathisia (inability to sit), anxiety, altered speech (difficult with speech), severe dizziness, syncope (fainting), parageusia (a bad taste in the mouth), tinnitus (ears ringing), blurred vision, tremors (an involuntary quivering movement, muscle spasms (twitching), depression, fatigue (a state of mental and/or physical weakness), nausea, chills, miosis (constriction of the pupil), angina (chest pain), tachycardia (fast heart rate), arrhythmia (irregular heartbeat), sternutation (sneezing), hyperhidrosis (increases sweating), arthralgia (joint pain), joint rigidity (stiffness), change in balance

Severe: Paresthesia (tingling or prickling, "pins and needles"), extremity edema (swelling of the arms and legs due to fluid), asthenia (abnormal physical weakness or lack of energy), wheezing (chest tightness), fever, itching, bad cough, blue skin color, seizures, swelling of face, lips, tongue or throat.

## Possible risks of Bupivacaine - Liposomal Bupivacaine (Exparel®):

Mild: Headache, insomnia (inability to fall asleep), muscle spasms (twitching), or back pain.

Moderate: Akathisia (inability to sit), anxiety, altered speech (difficulty with speech), severe dizziness, syncope (fainting), parageusia (a bad taste in the mouth), tinnitus (ears ringing), blurred vision, tremors (an involuntary quivering movement, muscle spasms

IRB – 16-1571 Consent Version 3/23/2020

(twitching), depression, fatigue (a state of mental and/or physical weakness), nausea, chills, miosis (constriction of the pupil), angina (chest pain), tachycardia (fast heart rate), arrhythmia (irregular heartbeat), sternutation (sneezing), hyperhidrosis (increased sweating), arthralgia (joint pain), joint rigidity (stiffness), change in balance.

Severe: Paresthesia (tingling or prickling, "pins and needles"), extremity edema (swelling of the arms and legs due to fluid), asthenia (abnormal physical weakness or lack of energy), wheezing (chest tightness), fever, itching, bad cough, blue skin color, seizures, swelling of face, lips, tongue or throat.

#### 4. BENEFITS

## What are possible benefits of participating in the research?

Participation in this study may help to improve your pain control after surgery, but it is also possible that your condition may worsen. There is no guarantee that you will personally benefit by participating in this research study. Your participation in this study may provide information that may help other people undergoing similar surgery in the future.

#### 5. COSTS

### Are there any costs to you if you participate in this study?

The following research study services are being done only because you are participating in this research study and will be paid for by the study sponsor and will not be billed to you or your health insurance plan. These "research only" services include: liposomal Bupivacaine (Exparel®).

Your surgery and post-operative care are standard of care and considered to be conventional routine clinical services that you would have received even if you were not participating in the research study. These will be billed to you or your health insurance plan. Examples of these routine services include: bupivacaine, your hospital stay, drugs used to control your pain after your operation, routine tests and services. You are responsible for paying any deductibles, copayments or co-insurance that are a normal part of your health insurance plan.

#### 6. COMPENSATION

## Are there any payments to you if you participate in this study?

There is no compensation for participation in this study.

Medications under investigation in this study already have approval by the Food and Drug Administration (FDA) for administration to achieve post-operative analgesia and

IRB – 16-1571 Consent Version 3/23/2020

are currently available as a prescription medication to licensed medical providers. There is no opportunity for commercialization.

#### 7. RESEARCH RELATED INJURY

# What will happen if you are injured as a result of taking part in the research?

In the event you are injured as a result of participation in this research, medical care is available to you. The costs of such medical care will be billed to you or your insurance company. There are no plans to provide compensation for lost wages, direct or indirect losses. The Cleveland Clinic will not voluntarily provide compensation for research related injury. You are not waiving any legal rights by signing this form. Further information about research related injury is available by contacting the Institutional Review Board at (216) 444-2924.

#### 8. PRIVACY AND CONFIDENTIALITY

# What will happen to your information that is collected for this research?

Cleveland Clinic has rules and procedures to protect information about you. Federal and State laws also protect your privacy.

The research team working on the study will collect information about you. This includes your health information, data collected for this research study and personal identifying information including your name, address, date of birth and other identifying information.

Generally, only people on the research team will know your identity and that you are in the research study. However, sometimes other people at Cleveland Clinic may see or give out your information. These include people who review research studies including the Institutional Review Board and Research Compliance, their staff, lawyers, or other Cleveland Clinic staff.

People outside Cleveland Clinic may need to see your information for this study. Examples include government groups (such as the Food and Drug Administration), safety monitors, other hospitals in the study and the sponsor of the research and their agents. Cleveland Clinic will do our best to ensure your information is kept confidential and that only the health information which is minimally required to conduct the study is used or disclosed to people outside Cleveland Clinic; however, people outside Cleveland Clinic who receive your information may not be covered by this promise.

You do not have to give this permission to use and give out your information; however you will not be able to participate in this research study without providing this permission by signing this consent form. The use and disclosure of your information has no expiration date.

IRB – 16-1571 Consent Version 3/23/2020

You may cancel your permission to use and disclose your information at any time by notifying the Principal Investigator in writing, insert name and address of the PI. If you do cancel your permission to use and disclose your information, your participation in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in the study.

Part of this study involves questionnaires. There are no physical risks associated with this portion of the study. Some of the questions asked as part of the study, may make you feel uncomfortable. You may refuse to answer any of the questions. There is a potential risk of loss of confidentiality of your data. Every effort will be made to keep your information confidential through the use of the following safeguards. Study information will be stored in a manner compliant with the Health Insurance Portability and Accountability Act (HIPAA) within the Cleveland Clinic. This includes storage on password protected computers owned and managed by the Cleveland Clinic. Only authorized individuals will have access, co-investigators will need to sign separate addenda acknowledging their review of this IRB application, and affirm adherence to the same policies.

## 9. QUESTIONS

### Who Do You Call With Questions Or Problems?

If you have any questions, concerns or complaints about the research, or develop a research-related problem, contact Dr. John Rodriguez at (216) 444-6664. If you have any questions after hours please call the general surgery resident on call at (216) 444-2000 or (800) 223-2273. If you have questions about your rights as a research subject, you should contact the Institutional Review Board at (216) 444-2924.

#### 10. VOLUNTARY PARTICIPATION

#### What are your rights as a research participant?

Taking part in this study is voluntary. You will be told of any new, relevant information from the research that may affect your health, welfare, or willingness to continue in this study. You may choose not to take part or may leave the study at any time. Withdrawing from the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to withdraw from the study you should discuss with your study doctor your decision to ensure a safe withdrawal.

IRB – 16-1571 Consent Version 3/23/2020

## 11. SIGNATURES

# **Statement of Participant**

I have read and have had verbally explained to me the above information and have had all my questions answered to my satisfaction. I understand that my participation is voluntary and that I may stop my participation in the study at any time. Signing this form does not waive any of my legal rights. I understand that a copy of this consent will be provided to me. By signing below, I agree to take part in this research study.

| Printed name of Participant | | |
|---|---|---|
| Signature of Participant | Date | |
| Statement of Person Conducting Int | ormed Consent Discussion | |
| | nined in this document with the participan tands the risks, benefits, alternatives and a study. | t and it is |
| Printed name of person obtaining cons | ent | |
| Signature of person obtaining consent | Date | |

